CLINICAL TRIAL: NCT03934359
Title: A Phase Ⅰ, Multi-Center, Open-Label Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Antitumor Activity of DN1508052-01 as a Single Agent When Administered Subcutaneously to Adult Patients With Advanced Solid Tumors
Brief Title: A Study to Evaluate the Safety, Tolerability of DN1508052-01 in Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai De Novo Pharmatech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DN1508052-01-101
Record Dates: First submitted 2019-04-28; First posted 2019-05-01 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Intervention Model Description: A phase Ⅰ,multi-center, open-label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: DN1508052-01 — DN1508052-01 will be administered subcutaneously on Day 1, Day 8 and Day 15 of each cycle.

SUMMARY:
This is a phase I, open-label, multicenter study in adult patients with advanced solid tumors that have progressed despite standard therapy or for which no standard therapy exists. DN1508052-01 will be administered subcutaneously on Day 1, Day 8 and Day 15 in 28-day cycles. Other dose regimens may be explored based on the analysis of emerging PK, pharmacodynamics (PD) and safety data. This study is designed to determine the MTD, RP2D and investigate the safety, tolerability, PK, biomarkers, HPV status and ISR in DN1508052-01-treated patients.

DETAILED DESCRIPTION:
Study Population is adult patients (≥18 years) with histologically or cytologically confirmed, unresectable advanced solid tumors that have progressed despite standard therapy or for which no standard therapy exists.The selected starting dose, 0.01 mg/m2 of DN1508052-01, SC, on Day 1, Day 8 and Day 15 of each cycle.The starting dose will proceed with one patient. The next dose 0.1 mg/m2 will be explored if safety data permit in that there is no instance of a ≥ Common Terminology Criteria for Adverse Event (CTCAE v5.0) Grade 2 AE that is at least possibly related to the study intervention.then Dose escalation will then proceed following the 3+3 cohorts design.Dose escalation will continue until MTD or RP2D is reached, or the dose escalation will be terminated at the discretion of Investigators and Sponsor (or its designee) based on the analyses of emerging PK, PD, safety and efficacy data.The Primary objective is to determine the maximum tolerated dose (MTD) and recommended phase Ⅱ dose (RP2D) and assess dose-limiting toxicity (DLT) of DN1508052-01 as a single agent when administered subcutaneously to adult patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older;
2. Patients with histologically or cytologically confirmed, unresectable advanced solid tumors that have progressed despite standard therapy or for which no standard therapy exists;
3. Patients must have at least one measurable lesion as defined by RECIST v1.1;
4. ECOG performance score 0 or 1;
5. Life expectancy ≥ 3 months;
6. Patients who have sufficient Baseline organ function and whose laboratory data meet the following criteria at enrollment:

   1. Absolute neutrophil count （ANC）≥1.5 × 109/L;
   2. Platelets ≥100 × 109/L;
   3. Hemoglobin ≥90g/dL;
   4. Liver function:

      Serum bilirubin ≤1.5 × upper limit of normal (ULN) or ≤ 3×ULN in any subject with Gilbert's Syndrome; Aspartate aminotransferase（AST） and alanine aminotransferase（ALT） ≤2.5 × ULN without liver metastases, or ≤5 × ULN if the patient has documented liver metastases;
   5. International normalization ratio ≤1.2 if the patient is not on anticoagulants, or ≤3 if the patient is on anticoagulants;
   6. Serum creatinine ≤1.5 mg/dL, or estimated glomerular filtration rate (eGFR)≥60 mL/min/1.73 m2;
7. Women of childbearing potential must have a negative serum pregnancy test prior to study entry, and agree to use adequate contraception from study entry through at least 1 month after the last dose of study drug. A female patient of nonchildbearing potential will have had at least 12 continuous months of natural (spontaneous) amenorrhea, follicle stimulating hormone level ≥40 mIU/mL at Screening, and an appropriate clinical profile (e.g., age appropriate, history of vasomotor symptoms), or have had surgical bilateral oophorectomy, hysterectomy, or tubal ligation ≥6 weeks prior to Screening; in the case of oophorectomy alone, reproductive status will be confirmed by hormone level assessment;
8. A male patient must agree to use adequate contraception (male condom with spermicide or provide evidence of successful vasectomy; sterile sexual partner; or female sexual partner who uses an intrauterine device with spermicide, a female condom with spermicide, a contraceptive sponge with spermicide, an intravaginal system, a double diaphragm with spermicide, a cervical cap with spermicide) from study entry through at least 1 month after the last dose of study drug;
9. Patients must provide written informed consent prior to any study procedures.

Exclusion Criteria:

* Disease

  1. Patients with symptomatic central nervous system (CNS) metastases or carcinomatous meningitis; Note: Patients with treated CNS metastases may participate in this trial if the patient has completed radiotherapy or surgery for CNS metastases >2 weeks prior to study entry and if the patient is neurologically stable ≥ 2 weeks (no new neurologic deficits from brain metastasis on Screening clinical examination, no new findings on CNS imaging, and no corticosteroids being used).

     Medical Conditions
  2. Patients who have a history of another primary malignancy, with the exception of locally excised non-melanoma skin cancer and carcinoma in situ of uterine cervix. A patient who has had no evidence of disease from another primary cancer for 3 or more years is allowed to participate in the study;
  3. Patients who have a known history of active hepatitis C or chronic hepatitis B ("active hepatitis" defined as HCV RNA level ≥ 103 copies/mL for hepatitis C or HBV DNA level ≥ 104 copies/mL for hepatitis B at Screening);
  4. Patients who have a known diagnosis of human immunodeficiency virus (HIV);
  5. Patients who have any severe and/or uncontrolled medical conditions or other conditions that, in the opinion of the Investigator and Sponsor, could affect the patient's participation in the study such as:

     1. Uncontrolled diabetes mellitus, HbA1c≥8%;
     2. Malignant illnesses that are uncontrolled or whose control may be jeopardized by treatment with this study treatment;
     3. Moderate or severe hepatic impairment, i.e., Child-Pugh class B or C (see appendix 8.6);
     4. Autoimmune disorders with systemic therapy;
  6. Patients who with an allo-transplant of any kind (including those with a xenograft heart valve);
  7. Any significant ophthalmologic abnormality, including but not limited to the following:

     1. Grade 2 or greater severity syndrome of dry eye;
     2. Keratoconjunctivitis sicca;
     3. Sjogren's syndrome;
     4. Iritis;
  8. Patients who have a history of definite neurological disorders that affected brain function activity, including epilepsy or dementia;
  9. Active infections requiring antibiotic intravenous therapy at Screening;
  10. Pregnancy or lactation;
  11. Patients with any comorbid medical disorder that, in the opinion of the Investigator or Sponsor, may increase the risk of toxicity; Organ Function and Laboratory Values
  12. Patients who have impaired cardiac function or clinically significant cardiac diseases, including any of the following:

      1. Baseline QT interval corrected for heart rate using Fridericia's formula >480 msec or congenital long QT syndrome;
      2. Concomitant diseases that could prolong the QT interval, as assessed by the Investigator, such as autonomic neuropathy (caused by diabetes or Parkinson's disease), cirrhosis, uncontrolled hypothyroidism, or grade 3 or greater severity electrolyte abnormality (CTCAE v5.0);
      3. Concomitant medications known to prolong the QT interval;
      4. History or presence of serious uncontrolled ventricular arrhythmias;
      5. Left ventricular ejection fraction <50% assessed by echocardiogram;
      6. Any of the following within 3 months prior to the first dose of study medication: myocardial infarction, severe/unstable angina, coronary artery bypass graft, congestive heart failure, cerebrovascular accident, or transient ischemic attack;
      7. Other clinically significant heart disease such as congestive heart failure NYHA Class Ⅱ or greater severity and requiring heart transplant or uncontrolled hypertension (systolic blood pressure > 150 mmHg or diastolic blood pressure > 100 mmHg, in spite of antihypertensive medication); Prior Therapy
  13. Chemotherapy, biologic therapy, herbal therapy, radiotherapy or investigational agents within 5 half lives or within 4 weeks (whichever is longer) prior to administration of the first dose of study drug on Day 1 or have not recovered to grade 1 or below from the side effects of such therapy (excluding cases of alopecia);
  14. Patients received potent CYP3A4 inducer or inhibitor within 2 weeks prior to administration of the first dose of study drug on Day 1.
  15. Patients received systemic corticosteroids within 2 weeks prior to administration of the first dose of study drug on Day 1.
  16. Major surgery for any cause within 4 weeks of first dosing;
  17. Treated with immunomodulator (e.g., motolimod, GS9688, IMO4200, E-6742, E-6887, etc).
  18. Patients who have a history of allergic reactions (significant urticaria, angioedema, anaphylaxis) attributed to compounds of similar chemical or biologic composition to DN1508052-01; Patients with scheduled surgeries or who are, in the Investigator's opinion, likely to require surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-09-18 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
the maximum tolerated dose (MTD) | 28 days
  MTD is the highest dose of DN1508052-01 in subjects with DLT less than 33.3% during the DLT observation in the dose escalation

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Up to 24 months
  Assessment of the cidence and severity of treatment-related AEs in who received at least 1 dose of in DN1508052-01
Time to peak (Tmax) of plasma concentration | Up to 2 months
  Pharmacokinetics profile of DN1508052-01 :Time to peak (Tmax) of plasma concentration
Maximum plasma concentration (Cmax) | Up to 2 months
  Pharmacokinetics profile of DN1508052-01 : Maximum plasma concentration (Cmax)
Halflife (T1/2) | Up to 2 months
  Pharmacokinetics profile of DN1508052-01 : Halflife (T1/2)
Clearance/ bioavailability (CL/F) | Up to 2 months
  Pharmacokinetics profile of DN1508052-01 : Clearance/ bioavailability (CL/F)
Area under curve (AUC) | Up to 2 months
  Pharmacokinetics profile of DN1508052-01 : Area under curve (AUC)
Efficacy Assessments | Up to 24 months
  Subjects will be assessed using RECIST v1.1. The primary aim is to demonstrate clinically meaning in ORR

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of California San Diego-Moores Cancer Center, La Jolla, California
  - Washington University School of Medicine - Siteman Cancer Center, St Louis, Missouri
  - University of Washington - Seattle Cancer Care Alliance, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No